CLINICAL TRIAL: NCT02329288
Title: Retrobulbar Triamcinolone Acetonide Injection in the Treatment of Nonarteritic Anterior Ischemic Optic Neuropathy
Brief Title: Retrobulbar Triamcinolone Acetonide Injection in the Treatment of NA-AION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, pandongyan, M.D., Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SecondMMU2014
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Triamcinolone Acetonide; Optic Neuropathy, Ischemic
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triamcinolone Acetonide (Active Comparator): 40mg/1ml
  Interventions: Drug: Triamcinolone Acetonide
- placebo (Placebo Comparator): 1ml
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Triamcinolone Acetonide
  Arms: Triamcinolone Acetonide
Drug: placebo
  Arms: placebo

SUMMARY:
NAION produces an ischemic insult in the optic nerve head presumably due to the hypoperfusion of the short ciliary arteries that supply it.

Intravenous injection of glucocorticoid have proven to be effective in treatment of Nonarteritic Anterior Ischemic Optic Neuropathy,but have some side effects. the investigators believe that offering them Retrobulbar Triamcinolone Acetonide Injection that might halt the progression of the visual acuity and visual field loss if our hypothesis is correct, would greatly improve their chances of avoiding blindness.

ELIGIBILITY:
Inclusion Criteria:

Sudden mono ocular vision loss associated with optic disc edema and positive Marcus Gunn (<30 days)

Exclusion Criteria:

Any eye disease except NAION(Nonarteritic Anterior Ischemic Optic Neuropathy) Neurologic defect Abnormal ESR, CRP, any history of retina or vitreal surgery Severe corneal opacity which makes retina examination impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Best corrected visual acuity(BCVA) | baseline and 1month, 3month

SECONDARY OUTCOMES:
Changes of Visual Field | baseline and 1month, 3month

CONTACTS AND LOCATIONS:
Overall Officials: shihong zhao, Study Director — department of ophthalmology